CLINICAL TRIAL: NCT05363176
Title: Telehealth CBT to Increase Engagement in Pain Treatment Among Veterans Using Prescription Opioids
Brief Title: Treatment, Pain, and Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDR 21-018
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Prescription opioids; Treatment; Treatment engagement; Beliefs
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two interventions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessors will not know what condition that the participant was allocated to, nor will the statistician who is one of the co-investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT for Treatment Seeking (Experimental): CBT delivered over the course of 1, ~45 minute session delivered via telehealth.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Treatment Seeking
- Pain Treatment Education (Active Comparator): Pain treatment education is delivered over the course of 1, ~45 minute session delivered via telehealth
  Interventions: Behavioral: Pain treatment education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Treatment Seeking — CBT delivered over the course of 1, ~45 minute sessions delivered via telehealth.
  Other Names: CBT-TS
  Arms: CBT for Treatment Seeking
Behavioral: Pain treatment education — Pain treatment education describes a variety of pain treatments offered in the VA. It is delivered over the course of 1, ~45 minute session delivered via telehealth
  Arms: Pain Treatment Education

SUMMARY:
Background: Chronic pain and negative consequences of long-term opioid therapy are related public health concerns associated with significant functional impairment, high psychiatric comorbidity, and premature mortality, particularly among Veterans. Clinical Practice Guidelines for opioid prescribing and pain management recommend using non-pharmacological approaches as first-line treatments. Psychosocial interventions (e.g., cognitive-behavioral therapy) have strong evidence supporting their ability to improve pain outcomes. Patient beliefs about the stigma associated with psychological interventions, opioid analgesics, ability of psychosocial intervention to improve pain among others can greatly interfere with the patients' ability to initiate and maintain engagement in psychosocial interventions and other non-pharmacological approaches.

Significance/Impact: Without a concerted effort at affecting beliefs that impede engagement in treatment, Veterans who may benefit from the treatment, will not receive it. This can result in continued risk for negative consequences associated with long-term opioid therapy and inadequate pain management. Cognitive-Behavioral Therapy for Treatment Seeking (CBT-TS) is an evidence-based intervention that directly intervenes on beliefs that act as barriers to treatment initiation and retention. By intervening on these beliefs, this study has the potential to improve engagement in psychosocial pain interventions and other non-pharmacological pain treatments, which will improve pain-related interference and functioning and reduce reliance on opioid analgesics. This study addresses VHA/VA Veteran care priorities including opioid use, pain management, and access and directly addresses priorities of the HSR&D Targeted Solicitation for Service Directed Research on Opioid Safety and Opioid Use Disorder.

Innovation: The proposed study is the first application of CBT-TS for Veterans with chronic pain who are receiving opioid analgesics-a notably high-risk, treatment-resistant population. This is the first study to directly intervene on thoughts about psychosocial interventions.

Specific Aims: The specific aims are to: test the effects of CBT-TS to increase initiation of psychosocial interventions for pain among Veterans receiving opioid analgesics for chronic pain (Aim 1), test the effects of CBT-TS to increase the retention in psychosocial interventions for pain among Veterans receiving opioid analgesics for chronic pain (Aim 2), and evaluate the effects of CBT-TS in improving pain and substance use outcomes among Veterans receiving opioid analgesics for chronic pain (Aim 3). The investigators will also test the effects of CBT-TS on the initiation of and retention to other non-pharmacological pain treatments (Exploratory Aim).

Methodology: Participants (N = 300) will be randomized to either the CBT-TS condition or an education control condition. Participants in both conditions will complete assessments on pain, treatment engagement, and opioid use at baseline, and 1-, 3-, and 6-months post-treatment to assess primary, secondary, and exploratory outcomes.

Implementation/Next Steps: Results from this study will provide critical information on increasing engagement of psychosocial interventions for pain, which can be used to inform future implementation and dissemination efforts. The research team will work with the VHA National Pain Management and Opioid Safety office and the VHA Office of Patient Centered Care & Cultural Transformation to identify implementation and dissemination efforts. CBT-TS is undergoing current implementation research to increase mental health functioning and this effort could be expanded to also increase treatment engagement of psychosocial interventions for pain and other non-pharmacological pain treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include English-speaking Veterans on long-term opioid therapy prescribed opioid analgesics (>20mg morphine equivalent daily [MEDD] and at least a 90 days supply).
* Participants must report pain that occurs on at least half the days for six months.

  * They must score at least a 4 on each item of the three items on a brief pain intensity and interference measure.

Exclusion Criteria:

* Veterans will be excluded if they are currently undergoing oncology treatment, are hospice patients, and have a recent or upcoming surgery.
* Veterans will be excluded if they are currently engaged (i.e., within the past month) in non-pharmacological pain treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Medical Record Review and Treatment Utilization Form | Baseline to 6-months post-treatment
  This will capture treatment initiation and treatment retention information including treatment types, dates of service, number of sessions, and type and dose of VHA and non-VHA medications dispensed.

SECONDARY OUTCOMES:
Pain Treatment Willingness Scale (PTWS) | Baseline to 6-months post-treatment
  Beliefs about psychosocial and other non-pharmacological pain treatments will be assessed using a modified PTWS. The scale consists of seven items assessing respondents' willingness to use opioids or non-pharmacological approaches using a 6-point rating scale. (1 = "not at all willing" to 6 "extremely willing").
Medication Beliefs Questionnaire | Baseline to 6-months post-treatment
  The MBQ uses five items to assess beliefs about one's response to, relief from, and potential for addiction to opioid analgesics. Respondents are asked to select one of five responses for each item (e.g., "None at all" to "Complete", "Much worse" to "Much better").
Beck Hopelessness Scale (BHS) | Baseline to 6-months post-treatment
  The BHS contains 20 true-false items designed to assess beliefs about the future. Higher scores represents greater hopelessness.
Pain Catastrophizing Scale | Baseline to 6-months post-treatment
  The PCS is a 13-item measure, with each item rated on a 5-point rating scale (0 = "Not at all" to 4 = "All the time"). Higher scores represent more rumination, magnification, and helplessness over pain.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline to 6-months post-treatment
  The PSEQ is an 11-item measure that assesses one's confidence in performing activities while in pain.
Tampa Scale for Kinesiophobia-11 (TSK-11) | Baseline to 6-months post-treatment
  The TSK-11 is an 11-item measure assessing pain-related fear of movement or injury with higher scores representing greater fear of movement.

OTHER OUTCOMES:
PROMIS Profile-29 | Baseline to 6-months post-treatment
  The PROMIS-29 provides a profile of one's health-related quality of life with components including pain interference, physical functioning, sleep disturbance, social functioning, anxiety, fatigue, and depression.
Opioid use | Baseline to 6-months post-treatment
  A 17-item measure will be used that assesses the frequency of aberrant drug-related behaviors and other behaviors that are prevalent among pain patients who are using prescription opioids. The rating scale ranges from 0 ("Never") to 4 ("Very Often"), with higher scores indicating greater risk.

CONTACTS AND LOCATIONS:
Overall Officials: Lisham Ashrafioun, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05363176/ICF_000.pdf